CLINICAL TRIAL: NCT01692288
Title: Evaluation of the Effectiveness of the First Born® Program for New Parents in Santa Fe County, New Mexico
Brief Title: Evaluation of the Effectiveness of a Home Visiting Program for New Parents in New Mexico
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Responsible Party: Principal Investigator, Rebecca Kilburn, Senior Economist, RAND
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K7051-07-03
Record Dates: First submitted 2012-09-14; First posted 2012-09-25 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Infant Health Risk Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Offered First Born® Program services (Experimental): Family and first-born child are selected to be offered First Born® Program home visiting services.
  Interventions: Behavioral: First Born® Program home visiting services
- Not offered First Born® Program services (No Intervention): Family and first-born child are not selected to be offered First Born® Program home visiting services.

INTERVENTIONS:
Behavioral: First Born® Program home visiting services — Family and first-born child are offered and/or receive weekly First Born® Program home visiting services between pregnancy and the child's third birthday. Families are eligible to enroll in the program from pregnancy up to two months after birth.
  Arms: Offered First Born® Program services

SUMMARY:
The purpose of this study is to determine if children and mothers who participate in the First Born® Program (FBP) experience better outcomes than they would have in the absence of the program. The evaluation employs a randomized trial design to assess the effectiveness of the FBP in the Santa Fe County, NM, site. FBP is a home visitation program that uses clinically trained professionals to provide first-time parents with information, training, and access to resources designed to promote early childhood development. Services are free and may begin at any time during pregnancy or up to two months after the baby's birth and may continue until the child is three years old. In addition, a nurse postpartum home visit is offered to the parents of all participating newborns. The FBP model builds on other home visiting and prevention programs that have been shown to improve long-term outcomes of children and their families.

ELIGIBILITY:
Inclusion Criteria:

* First-time parent
* Mother is currently pregnant or child is less than two months old
* Lives within Santa Fe County, New Mexico
* Parent accepts referral to First Born Program

Exclusion Criteria:

* Child is not first born
* First-born child is two months or older
* Parent resides outside Santa Fe County
* Parent has not been referred to First Born Program

Max Age: 2 Months | Sex: All
Age Groups: Child
Enrollment: 278 (Actual)
Dates: Start 2012-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with child health or development risk factors | First year of life

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Kilburn, PhD, Principal Investigator — RAND
Locations (1):
- United Way of Santa Fe County First Born® Program, Santa Fe, New Mexico, United States

REFERENCES:
- [Background] Kilburn MR, Cannon JS. Home Visiting Start-Up: Lessons Learned From Program Replication in New Mexico. J Prim Prev. 2015 Aug;36(4):275-9. doi: 10.1007/s10935-015-0392-5. PMID 25921835
- [Background] Kilburn, M.R. Lessons from the randomized trial evaluation of a new parent program: when the evaluators see the glass as half full, and the community sees the glass as half empty. J Exp Criminol (2012) 8: 255. doi:10.1007/s11292-012-9152-1
- [Result] Kilburn MR, Cannon JS. Home Visiting and Use of Infant Health Care: A Randomized Clinical Trial. Pediatrics. 2017 Jan;139(1):e20161274. doi: 10.1542/peds.2016-1274. Epub 2016 Dec 15. PMID 27980028